CLINICAL TRIAL: NCT05845216
Title: Effect of Transcranial Near InfraRed Light on Cerebral Function in Young and Healthy Older Subjects: a Functional Magnetic Resonance Imaging (fMRI) Study (TIROC)
Brief Title: Effect of Transcranial Near InfraRed Light on Cerebral Function in Young and Healthy Older Subjects: a FMRI Study (TIROC)
Acronym: TIROC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Commissariat A L'energie Atomique (Other Government); Fonds de Dotation Clinatec (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 38RC22.0227
Record Dates: First submitted 2023-03-15; First posted 2023-05-06 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Healthy Volunteers
Keywords: Transcranial photobiomodulation; near InfraRed; fMRI; brain function

STUDY DESIGN:
Intervention Model Description: The Primary Purpose of this clinical trial is to test a prototype device for feasibility and not health outcomes. This study is conducted to confirm the design and operating specifications of a device before beginning a full clinical trial.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ACTIVE tPBM (Experimental): one session of 24-min tPBM with the active device (tPBM helmet with 80 Light-Emitting Diodes (LEDs) emitting red and near-infrared light at 670 - 810nm)
  Interventions: Device: ACTIVE Transcranial photobiomodulation (tPBM)
- SHAM tPBM (Sham Comparator): one session of 24-tPBM with a sham device visually identical to the active device
  Interventions: Device: SHAM Transcranial photobiomodulation (tPBM)

INTERVENTIONS:
Device: ACTIVE Transcranial photobiomodulation (tPBM) — fMRI records before and after ACTIVE Transcranial photobiomodulation (tPBM)
  Arms: ACTIVE tPBM
Device: SHAM Transcranial photobiomodulation (tPBM) — fMRI records before and after SHAM Transcranial photobiomodulation (tPBM)
  Arms: SHAM tPBM

SUMMARY:
Numerous studies have shown that the extra-cranial application of near infrared light (λ=600-1000nm) (also called transcranial photobiomodulation or tPBM), has a positive impact on brain function in both humans and experimental animal models and a neuroprotective effect in animal models. Several of these studies have reported that tPBM could impart more beneficial effects in aged or diseased brains. The primary objective of this study is to use fMRI to compare the cerebral activations in response to a finger tapping motor task, before and after 24min of tPBM versus sham stimulation, in old and young healthy human subjects.

The hypothesis of the investigators is that tPBM improves brain function in participants who will be treated using the active device in comparison with those treated with the sham device and that this effect should will be more pronounced in the older subjects.

DETAILED DESCRIPTION:
Many studies have shown that the extra-cranial application of light in the red and near infrared range (λ=600-1000nm), also called transcranial PhotoBioModulation (tPBM), could have a neuroprotective effect and a positive impact on brain function in the mammalian brain.

At the cellular level, it is thought that the mechanism mainly relies on the activation of the cytochrome C oxidase and/or interfacial nanowater, two photoacceptors located within the mitochondria that absorb red and near infrared photons. The interaction between the photons and the photoacceptor results in a cascade of secondary events, activating the respiratory chain and increasing Adenosine TriPhosphate (ATP) synthesis, the main source of energy in the cell.

In humans, an increasing number of studies have reported an improvement of cognitive functions after one or several tPBM sessions in patients suffering Alzheimer's or Parkinson's disease, or in cases of stroke. Recently, some EEG and fMRI studies on healthy subjects, young and/or old, have also reported a modification of neuronal activation patterns at rest or during the performance of a cognitive task.

Regarding tPBM, this is a non-pharmacological and non-surgical treatment, for which no adverse effects have been reported. Further, the FDA has already approved the use of several PBM devices for therapeutic use in humans, for example, the treatment of pain, inflammation or dermal conditions.

Those preliminary results in humans are thus very encouraging. However, the precise mechanism of action remains to be better characterised, and further studies are required to better define its effects on the human brain and its indications for a therapeutic use. Moreover the extent tPBM influence on the brain of the elderly is still very unclear. In the present study, the investigators aim to evaluate brain function before and after a tPBM session, during the realisation of a motor task or at rest, while comparing a group of young and elderly subjects.

The working hypotheses of the investigators are as follows :

* tPBM will improve motor performances and brain function of all subjects, and to a greater extent that of the older subjects
* tPBM will change brain activity, reorganising large scale neuronal networks at rest.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman
* Aged 18 to 40 (young group), or 60 to 85 (elderly)
* Right-handed (Edinburgh score for hand laterality >70%)
* No taking psychoactive or anti-depressants medicine
* Normal or corrected vision
* Having expressed their consent to the research
* Affiliated to a social security scheme
* Registered in the national file of people lend themselves to biomedical research

Exclusion Criteria:

* Known cognitive disorder, neurologic trouble, neurodegenerative disease or psychiatric illness,
* Motor disorder able to impair the task management
* Contraindication for MRI (metallic implant, non-removable piercing, pace-maker, metallic prosthesis, claustrophobia , …)
* Montreal Cognitive Assessment (MoCA) score <26
* People referred to in Articles L1121-5 to L1121-8 of the Public Health Code(corresponds to all protected persons: pregnant, parturient or breastfeeding women, persons deprived of liberty by judicial or administrative decision, persons subject of psychiatric care, minors, and persons subject to a legal protection measure: guardianship, curators or safeguard of justice)
* Persons in period of exclusion from another clinical investigation
* Subjects participating in another clinic investigation,
* Subjects who would receive more than 4500 euros in compensation due to his participation in other biomedical research in the 12 months preceding this study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Cerebral activations in response to a Finger Tapping motor task. | 24 minutes
  Cerebral activation measured by fMRI (BOLD signal change) in response to a finger tapping motor tap (contrasted against a resting baseline), before and after tPBM/Sham stimulation

SECONDARY OUTCOMES:
Performances in the Finger Tapping motor task | 24 minutes
  Performances in the Finger Tapping motor task (correct movement execution speed) before and after tPBM / Sham stimulation
Functional connectivity (BOLD signal variations during the finger tapping task compared to rest state) | 24 minutes
  Functional connectivity measured by fMRI (BOLD signal variation during the Finger tapping task compared to rest state) before and after tPBM / sham stimulation

CONTACTS AND LOCATIONS:
Locations (1):
- Clinatec Cea/Chuga, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dole M, Auboiroux V, Langar L, Mitrofanis J. A systematic review of the effects of transcranial photobiomodulation on brain activity in humans. Rev Neurosci. 2023 Mar 17;34(6):671-693. doi: 10.1515/revneuro-2023-0003. Print 2023 Aug 28. PMID 36927734
- [Background] El Khoury H, Mitrofanis J, Henderson LA. Exploring the Effects of Near Infrared Light on Resting and Evoked Brain Activity in Humans Using Magnetic Resonance Imaging. Neuroscience. 2019 Dec 1;422:161-171. doi: 10.1016/j.neuroscience.2019.10.037. Epub 2019 Nov 1. PMID 31682952
- [Background] Dmochowski GM, Shereen AD, Berisha D, Dmochowski JP. Near-Infrared Light Increases Functional Connectivity with a Non-thermal Mechanism. Cereb Cortex Commun. 2020 Mar 19;1(1):tgaa004. doi: 10.1093/texcom/tgaa004. eCollection 2020. PMID 34296085
- [Background] Hamblin MR. Shining light on the head: Photobiomodulation for brain disorders. BBA Clin. 2016 Oct 1;6:113-124. doi: 10.1016/j.bbacli.2016.09.002. eCollection 2016 Dec. PMID 27752476
- [Background] Nizamutdinov D, Qi X, Berman MH, Dougal G, Dayawansa S, Wu E, Yi SS, Stevens AB, Huang JH. Transcranial Near Infrared Light Stimulations Improve Cognition in Patients with Dementia. Aging Dis. 2021 Jul 1;12(4):954-963. doi: 10.14336/AD.2021.0229. eCollection 2021 Jul. PMID 34221541